CLINICAL TRIAL: NCT01122082
Title: Influence of Respiratory Quotient on Food Liking, Food Wanting, Macronutrient Selection and Food Consumption in Humans
Brief Title: Respiratory Quotient and Food Liking, Food Wanting and Food Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Principal Investigator, Laurent BRONDEL, Professor, University of Burgundy
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: ABC123; CSGA-AA1234-01 (Registry Identifier: 02052009)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: energy intake; energy expenditure; macronutrient selection
MeSH Terms: conditions — Obesity | interventions — Eating; Metabolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: food preloads — Subjects will eat in the morning during breakfast 300g cottage cheese (627kJ - 147kcal; 13.2g carbohydrate, 0.3g fat, 23g protein) plus, according to the situations, either: 90g sucrose, HCB); 6g aspartame; 40g vegetable oil; 40g paraffin oil. Therefore two breakfast will have the same energy content (2072kJ - 495kcal), as did the other two(565 kJ - 135kcal).
  Other Names: food intake; metabolism

SUMMARY:
The purpose of this study is to observe the influence of carbohydrate-to-fat balance on liking, wanting and food consumption in humans.

16 normal-weight men (age: 23 ± 3 y)had completed a randomized 4-condition crossover study. The sessions differed by the composition of the breakfast which was rich in carbohydrates (HCB), low in carbohydrates (LCB), rich in fat (HFB) and low in fat (LFB). The HCB and HFB contained 2072 kJ, while the LCB and LFB contained 565 kJ. Two hours and 20 min later, energy expenditure (EE) and respiratory quotient (RQ) were measured before olfactory liking for 4 foods items and then ad libitum energy intake (EI) during a snack (sweet and fatty toast) were evaluated.

DETAILED DESCRIPTION:
In accordance with the carbohydrate-based models of feeding, one may expect that food choices as well as "liking" and "wanting" (the two components of the reward system) could be influenced by glycogen stores and the carbohydrate-to-fat balance. More precisely, one may expect that a high fat oxidation rate could increase liking and wanting carbohydrates to replenish glycogen stores and conversely, that a high carbohydrate oxidation rate could produce the reverse. In order to validate this hypothesis, the present study has been conducted to investigate in humans the influence of the carbohydrate-to-fat oxidation ratio on carbohydrate-to-fat selection and the food reward system.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Absence of medication
* Moderate physical activity (irregular and less than 5 h/wk)
* Low-smoking habit (less than 5 cigarettes/d)
* Normal body mass index (20< BMI <25)

Exclusion Criteria:

* Eating disorders
* Dieting or fasting
* Aversions for the foods offered and elevated 'cognitive restriction of eating' (score ≥ 7) according to the Three Factor Eating Questionnaire

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Respiratory quotient | 6 months
  Respiratory quotient is the ratio of CO2 production on oxygen consumption measured in the expiratory flow

SECONDARY OUTCOMES:
food liking | 6 months
  Food liking is the preference for 4 food items smelt
food wanting | 6 months
  food wanting is the selection of 4 kind of toasts during a snack
food consumption | 6 months
  is the amount of food eaten during the snack

CONTACTS AND LOCATIONS:
Overall Officials: Luc Penicaud, MD, Study Director — Centre National de la Recherche Scientifique, France
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brondel L, Landais L, Romer MA, Holley A, Penicaud L. Substrate oxidation influences liking, wanting, macronutrient selection, and consumption of food in humans. Am J Clin Nutr. 2011 Sep;94(3):775-83. doi: 10.3945/ajcn.111.017319. Epub 2011 Jul 27. PMID 21795442